CLINICAL TRIAL: NCT02174094
Title: Multi-site, Prospective, Randomised, Double-blind, Placebo-controlled, Parallel-group, Interventional Study to Evaluate the Efficacy, Safety, and Tolerability of Clobazam as Adjunctive Therapy in Paediatric Patients Aged ≥1 to ≤16 Years With Dravet Syndrome
Brief Title: Clobazam as Adjunctive Therapy in Paediatric Patients Aged ≥1 to ≤16 Years With Dravet Syndrome
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated due to recruitment challenges
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14362A
Record Dates: First submitted 2014-06-02; First posted 2014-06-25 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Dravet Syndrome
MeSH Terms: conditions — Epilepsies, Myoclonic | interventions — Clobazam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clobazam (Experimental): Clobazam - 1.0, 1.5 or 2.0 mg/kg/day (maximum 60 or 80 mg/day) twice daily (BID); Clobazam oral suspension 2.5 mg/mL, clobazam scored tablets 10 mg, orally
  Interventions: Drug: Clobazam
- Placebo (Placebo Comparator): Placebo to clobazam oral suspension 2.5 mg/mL and placebo to clobazam scored tablets 10 mg, orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clobazam
  Other Names: Onfi®
  Arms: Clobazam
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effect on the frequency of tonic-clonic and clonic seizures of clobazam as adjunctive therapy compared to placebo after 16 weeks of treatment in paediatric patients aged ≥1 to ≤16 years with Dravet Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Onset of seizures in the first year of life
* History of fever-induced prolonged seizures as determined by the Investigator
* These may include prolonged (approximately 15 minutes or longer) hemi-clonic seizures
* Multiple seizure types which may include:

  * generalised tonic-clonic (required for inclusion)
  * clonic (required for inclusion)
  * myoclonic jerks/seizures
  * history of normal development prior to seizure onset followed by development delay or regression after seizure onset
  * abnormal EEG consistent with Dravet Syndrome 2. The patient has a history of approximately 2 tonic-clonic or clonic seizures in 2 weeks 3. The patient is treated with at least 1 but no more than 3 antiepileptic drugs (AEDs) [Vagal Nerve Stimulator (VNS) and ketogenic diet will not be considered an AED] 4. Patient has at least 2 seizures during the Baseline Period of either 2 or 4 weeks

Exclusion Criteria:

1. The patient is taking stiripentol, verapamil, or felbatol. If patients have taken these drugs in the past, they need to have been off drug for 5 half-lives
2. The patient is taking a sodium channel blocker including, but not limited to, phenytoin, fosphenytoin, carbamazepine, oxcarbamazepine, lamotrigine, lacosamide, and rufinamide. If patients have taken these drugs in the past, they need to have been off drug for 5 half-lives
3. The patient is on cannabidiol, medical marijuana, or any drug that contains cannabinoids
4. The patient has received chronic treatment (≥2 weeks for any indication) with a benzodiazepine within at least 5 half-lives prior to screening. Rescue therapy for prolonged seizures is allowed
5. The patient has received clobazam within 3 months prior to the Screening Visit. If the patient has received clobazam in the past, discontinuation must not have been for adverse events or lack of efficacy

Other protocol-defined inclusion and exclusion criteria may apply.

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline to study completion/withdrawal in seizure rate for combined tonic-clonic and clonic seizure rates, based upon a calculation of seizure frequency determined from daily seizure diary counts | Baseline and from week 0 to week 16

SECONDARY OUTCOMES:
Percent change from baseline to study completion/withdrawal in seizure rate for combined tonic-clonic and clonic seizure rates, based upon a calculation of seizure frequency determined from daily seizure diary counts during 4 weeks of maintenance | Baseline and from week 4 to week 16
Percent change in seizure rate for myoclonic seizures determined from daily seizure diary counts | Baseline and from week 0 to week 16
Percent change in seizure rate for atypical absence seizures determined from daily seizure diary counts | Baseline and from week 0 to week 16
Percent change in seizure rate for complex partial seizures determined from daily seizure diary counts | Baseline and from week 0 to week 16
Percent change in seizure rate for all seizure types determined from daily seizure diary counts | Baseline and from week 0 to week 16
Number of initial treatment responders who returned to their baseline tonic-clonic and clonic seizure rate during the study (an assessment of tachyphylaxis) | Baseline and from week 0 to week 16
Percentage of initial treatment responders who returned to their baseline tonic-clonic and clonic seizure rate during the study (an assessment of tachyphylaxis) | Baseline and from week 0 to week 16
Percent change in seizure rate for myoclonic seizures determined from video EEG | Baseline and from week 0 to week 16
Percent change in seizure rate for atypical absence seizures determined from video EEG | Baseline and from week 0 to week 16
Change in Symptom and Seizure Activity Scale (Investigator and Parent/caregiver versions) | Baseline and from week 0 to week 16
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Up to Week 32
Columbia Suicide Severity Rating Scale (C-SSRS), categorisation based on Columbia Classification Algorithm of Suicide Assessment (C-CASA) categories (1, 2, 3, 4 and 7) for patients aged ≥ 6 years | Baseline and from week 0 to week 16
Number of Participants with Adverse Events of special interest as a Measure of Safety and Tolerability based on dose | Baseline and Week 32
Change in Vineland Adaptive Behaviour Scale (VABS) - all adaptive behavior sub-domains and maladaptive behaviors | Baseline and from week 0 to week 16

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (9):
- United States (8):
  - US010, Los Angeles, California
  - US001, Orlando, Florida
  - US003, Rochester, Minnesota
  - US005, Kansas City, Missouri
  - US0011, Dallas, Texas
  - US006, Dallas, Texas
  - US002, Houston, Texas
  - US004, Seattle, Washington
- MX003, Guadalajara, Mexico